CLINICAL TRIAL: NCT03268720
Title: Influence of the Immunosystem in Non-celiac Glutensensitivity
Acronym: NCGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, yurdagül zopf, Prof. Dr., University of Erlangen-Nürnberg Medical School
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: Glutensensitivity
Record Dates: First submitted 2017-08-15; First posted 2017-08-31 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Gluten Sensitivity
Keywords: gluten sensitivity; gluten-free diet; FODMAP diet; microbiome
MeSH Terms: conditions — Celiac Disease | interventions — FODMAP Diet; Diet, Gluten-Free

STUDY DESIGN:
Intervention Model Description: Participants consume a two week lasting low FODMAP diet, followed by 5 days washout, and subsequent two week gluten-free diet.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- healthy controls (Other): FODMAP low diet gluten-free diet
  Interventions: Other: FODMAP low diet; Other: gluten-free diet
- NCGS patients (Other): FODMAP low diet gluten-free diet
  Interventions: Other: FODMAP low diet; Other: gluten-free diet

INTERVENTIONS:
Other: FODMAP low diet — 2 week FODMAP low diet
Other: gluten-free diet — 2 week gluten-free diet

SUMMARY:
Patients with non-celiac gluten sensitivity (NCGS) complain about gastrointestinal and extraintestinal symptoms while consuming gluten-containing cereals. The symptoms strictly correlate with ingestion of gluten-containing cereals and disappear quickly under elimination diets. Till now, there are no specific markers to diagnose NCGS. This study aims to determine the effect of a low FODMAP diet (fermentable oligo-, di- and monosaccharides and polyols) and a glutenfree diet on the mucosal immunity, clinical symptoms, and psychological well-being. Furthermore, the influence of the diets on the microbiome will be analyzed.

DETAILED DESCRIPTION:
Patients with gluten-sensitivity are rigourously checked for wheat allergy and celiac disease. Genotyping for DQ2/8, serological detection of celiac specific antibodies, and gastroduodenoscopy are performed. Furthermore, a skin prick test and detection of wheat specific IgE are done.

After exclusion of celiac disease and wheat allergy patients are considered as patients with NCGS.

Patients and healthy controls are asked to consume a low FODMAP diet for two weeks, followed by a 5 day washout and subsequent two week gluten-free diet.

At the beginning and the end of each diet the participants fill in questionnaires concerning Nutrition (Freiburger Nutrition protocol), psychological well-being index (PGWB), gastrointestinal symptom Rating score (GSRS), and stool consistency (Bristol stool Chart). Furthermore, stool samples are selected at each time point to determine the microbial pattern.

NCGS patients with ongoing complaints will have a second gastroduodenoscopy at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* healthy controls
* patients with glutensensitivity

Exclusion Criteria:

* patients with glutensensitivity but without celiac disease or wheat allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Determination of clinical symptomatics | 2 weeks
  Analysis of the improvement of clinical symptoms according to gastrointestinal symptom Rating score
Determination of psychological symptoms | 2 weeks
  Improvement of well-being by questionnaire psychological General well-being index

SECONDARY OUTCOMES:
Nutrition Analysis for energy intake and nutritional composition by questionnaire Freiburger Nutrition protocol | 2 weeks
  Determination of nutrient intake according to questionnaire Freiburger Nutrition protocol. The questionnaire allows the detailed determination of energy intake, carbohydrates, fatty acids, and Protein.
Intraepithelial lymphocytes | 4 weeks
  numbers of intraepithelial lymphocytes in duodenal mucosa
Goblet cells | 4 weeks
  numbers of Goblet cells in duodenal mucosa
microbiome | 2 weeks
  Analysis of microbiota pattern

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine 1, Hector Center for Nutrition, Exercise and Sports, Friedrich-Alexander-University Erlangen-Nuremberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dieterich W, Schuppan D, Schink M, Schwappacher R, Wirtz S, Agaimy A, Neurath MF, Zopf Y. Influence of low FODMAP and gluten-free diets on disease activity and intestinal microbiota in patients with non-celiac gluten sensitivity. Clin Nutr. 2019 Apr;38(2):697-707. doi: 10.1016/j.clnu.2018.03.017. Epub 2018 Apr 4. PMID 29653862